CLINICAL TRIAL: NCT02474017
Title: An Open Study to Assess the Robustness of the CRC749 Device by Pharmaceutical Performance Following Twice Daily Dosing of MGR001 Administered Via Oral Inhalation in Subjects With Asthma or Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: An Open Study to Assess the Robustness of the CRC749 Inhaler
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharma UK Ltd. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGR001-1010; 2015-000463-13 (EudraCT Number)
Record Dates: First submitted 2015-06-03; First posted 2015-06-17 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Asthma; COPD
Keywords: Inhaler; Adolescent
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MGR001 (Experimental): MGR001 (FP/Salmeterol) (250/50 µg) twice daily (BID)
  Interventions: Drug: MGR001; Device: CRC749 inhaler

INTERVENTIONS:
Drug: MGR001 — Fluticasone Propionate / Salmeterol administered using CRC749 inhaler
Device: CRC749 inhaler

SUMMARY:
To confirm the robustness of the CRC749 inhaler.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 12 years of age.
2. A clinical diagnosis for at least 12 weeks prior to screening of asthma or COPD and stable treatment.
3. Spirometry following salbutamol showing FEV1 ≥40% of predicted normal and FEV1/FVC ratio <0.7 for COPD subjects.
4. Spirometry without salbutamol showing FEV1 ≥50% of predicted normal for asthma subjects.
5. Ability to use the CRC749 inhaler.

Exclusion Criteria:

1. Other chronic or active respiratory disorder or symptoms of, or treatment for a COPD or asthma exacerbation during the 28 days preceding screening.
2. History of long QT syndrome or screening ECG with QTcF greater than 480 milliseconds.
3. Current evidence of, or history within the 6 months prior to screening of unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, or myocardial infarction.
4. Subjects in whom Advair(R) Diskus(R) / Seretide(R) Accuhaler(R) are contra-indicated.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
In vitro Measurement of Emitted Dose | 3 Weeks
  CRC749 inhaler robustness will be assessed by in vitro testing of the CRC749 inhaler after 3 weeks of patient use of the MGR001 product.

SECONDARY OUTCOMES:
Adverse Events | 3 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard Allan, Study Director — Mylan Pharma UK Ltd.
Locations (2):
- United Kingdom (2):
  - Mylan Investigational Site, London
  - Mylan Investigational Site, Manchester

REFERENCES:
- [Derived] Allan R, Canham K, Wallace R, Singh D, Ward J, Cooper A, Newcomb C. Usability and Robustness of the Wixela Inhub Dry Powder Inhaler. J Aerosol Med Pulm Drug Deliv. 2021 Apr;34(2):134-145. doi: 10.1089/jamp.2020.1603. Epub 2020 Aug 31. PMID 32865454